CLINICAL TRIAL: NCT01908777
Title: A Phase 2 Multicenter Study of High Dose Chemotherapy With Autologous Stem Cell Transplant Followed by Maintenance Therapy With Romidepsin for the Treatment of T Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Washington (Other); Weill Medical College of Cornell University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-020
Record Dates: First submitted 2013-07-17; First posted 2013-07-26 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: T Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Drug Therapy; romidepsin; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high dose chemo w/asct + maintenance txt (Experimental): High dose chemotherapy (Carmustine), VP-16 (etoposide, Vepesid®), Cytarabine (Ara-C), Melphalan (Alkeran)with autologous stem cell transplant followed by maintenance therapy with Romidepsin (Istodax)
  Interventions: Other: High Dose Chemotherapy with Autologous Stem Cell Transplant Followed by Maintenance Therapy with Romidepsin

INTERVENTIONS:
Other: High Dose Chemotherapy with Autologous Stem Cell Transplant Followed by Maintenance Therapy with Romidepsin
  Other Names: Carmustine; VP-16 (etoposide, Vepesid®); Cytarabine (Ara-C); Melphalan (Alkeran); Romidepsin (Istodax)

SUMMARY:
The purpose of this study is to test the benefit of a chemotherapy drug called romidepsin in patients with T Cell Non-Hodgkin Lymphoma (T NHL) who have undergone autologous transplantation.

DETAILED DESCRIPTION:
The primary aim is to determine a preliminary estimate of the progression-free survival of patients with T NHL who receive maintenance romidepsin at 2 years post-transplant for patients transplanted in CR1 or PR1 with standard risk histologies.

Secondary aims include:

* Determine PFS at 2 yrs for patients transplanted in ≥CR/PR2 or for patients with high risk histologies.
* Determine the toxicities associated with romidepsin following autologous transplantation
* Determine the probability of OS at 2 years post transplant for all patients undergoing transplant
* Characterize the effect of romidepsin on immune recovery post HDT-ASCT
* OS and PFS 1 year after Romidespin completion

Patients who receive romidepsin after transplant will be evaluable for the primary endpoint, and will be counted towards the accrual total. Any patient who does not receive romidepsin after transplant, regardless of reason, will be replaced. We will also accrue a second cohort of 8 patients who are transplanted in >CR/PR2 and for high risk histologies to be analyzed for secondary endpoints only. This cohort will not be part of the primary endpoint and will be analyzed for summary statistics only. Patients who receive romidepsin after transplant will be counted towards the accrual total for Cohort 2. Any patient who does not receive romidepsin after transplant, regardless of reason, will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients over age 16 who are deemed eligible for transplant by their treating physician Disease status: CR or PR required. Remission status will be assessed at the completion of induction chemotherapy and prior to enrollment on protocol.

Diagnosis: The following histologies will need to be confirmed at MSK or locally for participating sites in order to be considered for HDT-ASCT and post-transplant maintenance romidepsin:

* PTCL
* AITL
* ALCL
* EaTCL
* Hepatosplenic Gamma Delta T cell lymphoma
* Adult T-cell leukemia/lymphoma
* Primary cutaneous gamma/delta T-cell lymphoma
* Extranodal NK/T-cell lymphoma, nasal type
* Primary cutaneous anaplastic large cell lymphoma
* Subcutaneous panniculitis-like T-cell lymphoma
* Mycosis fungoides/sezary syndrome Stem cell collection: A minimum of 2 x 106 CD34+ cells must have been collected

Laboratory test results within these ranges:

* Total bilirubin <= 1.5 x ULN
* AST (SGOT) and ALT (SGPT) <= 3 x ULN

Exclusion Criteria:

* Diagnosis: progressive disease at transplant work-up
* Prior therapy: prior autologous or allogeneic transplant
* Active and uncontrolled infection at time of transplantation including active infection with Aspergillus or other mold, or HIV infection
* Inadequate performance status/organ function defined by DLCO < 50% (adjusted for hgb), cardiac function as defined below, KPS < 60%.
* Pregnant or breast feeding. For males and females of child-producing potential, inability to use effective contraceptive methods during the study
* Prior therapy with romidepsin
* Central nervous system or meningeal involvement
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * QTc interval ≥ 500 milliseconds
  * Myocardial infarction within 6 months of transplantation. Subjects with a history of myocardial infarction between 6 and 12 months prior to transplant who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate
  * Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
  * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Appendix 1) In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix 2) and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD)
  * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes
  * Uncontrolled hypertension, defined as blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria
  * Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
  * Patients taking drugs leading to significant QT prolongation within the specified wash out period (See Appendix 3: Medications That May Cause QTc Prolongation).
  * Concomitant use of CYP3A4 inhibitors

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
The progression-free survival of patients | 2 Years
  The progression-free survival of patients with T NHL who receive maintenance romidepsin at 2 years post-transplant for patients transplanted in CR1 or PR1 with standard risk histologies.

SECONDARY OUTCOMES:
Progression Free Survival for patients with high risk histologies | 2 Years
  Determine PFS at 2 yrs for patients transplanted in ≥CR/PR2 or for patients with high risk histologies.
Toxicities | 2 years
  Determine the toxicities associated with romidepsin following autologous transplantation. Toxicities will be graded on a scale of 0 to 5 as described by the NCI- Common Terminology for Adverse Events (CTCAE), version 4.0
Probability of OS at 2 years post transplant | 2 year post transplant
  Determine the probability of OS at 2 years post transplant for all patients undergoing transplant
OS 1 year after Romidespin completion | 1 year
  OS 1 year after Romidespin completion
PFS 1 year after Romidespin completion | 1 year
  PFS 1 year after Romidespin completion

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Fred Hutchinson Cancer Research Center (Data Collection Only), Seattle, Washington
  - University of Washington (Data Collection Only), Seattle, Washington

REFERENCES:
- [Derived] Khan N, Dahi PB, Khimani F, Shustov AR, Shadman M, Ruan J, Moskowitz AJ, Zelenetz AD, Noy A, Straus DJ, Drullinsky P, Hamilton A, Kumar A, Sauter CS, Shah GL, Matasar MJ, Drill E, Davey T, Hancock H, Ganesan N, Galasso N, van Beisen K, Giralt S, Horwitz SM. Maintenance therapy with romidepsin after autologous stem-cell transplant for peripheral T-cell lymphoma. Blood Adv. 2025 Sep 23;9(18):4687-4692. doi: 10.1182/bloodadvances.2024014263. PMID 40179392
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/